CLINICAL TRIAL: NCT03553043
Title: Energy Labelling for Alcohol Drinks in New Zealand: Consumers Perceptions and Impacts on Purchase Behaviour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Collaborators: Te Hiringa Hauora/Health Promotion Agency (Unknown)
Responsible Party: Principal Investigator, Natalie Walker, Associate Professor, University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NI373821
Record Dates: First submitted 2018-05-20; First posted 2018-06-12 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Consumption, Alcohol; Drinking, Alcohol
Keywords: consumer behaviour; alcohol labelling; energy labelling
MeSH Terms: conditions — Alcohol Drinking | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned (1:1:1:1 ratio, stratified by ethnicity and alcohol use) by computer to view on-line one of four label conditions.
Masking Description: Due to the nature of the intervention, it will not be possible to blind participants or research staff to the different conditions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Energy Label 1 (Experimental): Alcoholic beverage displayed with Energy label 1
  Interventions: Behavioral: Intervention
- Energy Label 2 (Experimental): Alcoholic beverage displayed with Energy Label 2
  Interventions: Behavioral: Intervention
- Energy Label 3 (Experimental): Alcoholic beverage displayed with Energy Label 3
  Interventions: Behavioral: Intervention
- Unlabelled (Placebo Comparator): Alcohol beverage displayed unlabelled.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Intervention — Energy label condition.
  Arms: Energy Label 1; Energy Label 2; Energy Label 3
Behavioral: Control — No label
  Arms: Unlabelled

SUMMARY:
A two-stage qualitative and quantitative study to provide insight into consumers' awareness of energy in alcoholic beverages, and how energy labelling effects consumer behaviour.

DETAILED DESCRIPTION:
Rationale: In 2016/2017, one in five (19.5%) New Zealand adults (≥15 years and older) had an alcohol drinking pattern that carriers a risk of harming the drinker or another, and one in three (32.9%) young adults aged 18 to 24 years are hazardous drinkers. To reduce alcohol-related harm and help New Zealanders make positive decisions about their alcohol use, strategies are needed that not only inform them about health risks but also alter the environment they find themselves in on a daily basis. Unlike most packaged food products, alcoholic beverages are not required to present a statement of the composition of the product, such as amount of alcohol, energy or the nutrient content. It has been suggested that in the absence of this information, consumers of alcohol have no idea how much energy, alcohol or kilojoules they are consuming. Research indicates that nutrition labelling of food and non-alcoholic beverage products does impact consumer perceptions and product evaluations. A recent poll by Stuff showed that 83% of 3,300 New Zealanders indicated that they want to know what they are consuming and supported placement of ingredients and nutritional information on alcohol products.

Objectives: To provide insight into consumers' awareness of energy in alcoholic beverages, and in their views on energy labelling of alcoholic beverages. The project also aims to explore the effects of different types of energy labelling on consumers alcohol purchase behaviour.

Design: Two-staged qualitative and quantitative study.

* Qualitative stage: Focus groups.
* Quantitative stage: Four-arm randomised controlled trial. This qualitative stage aims to test the effects of three different types of alcohol energy labels on alcoholic beverages on (online) purchase behaviour, compared to a control (no label) condition, using an 'online shopping cart'.

Recruitment: Panel.

Sample size: Qualitative stage: n=36 (six focus groups with six people per group); Quantitative stage: n=600 (n=150 participants per experimental condition).

ELIGIBILITY:
Inclusion Criteria:

* are ≥18 years of age;
* having purchased and consumed at least one alcoholic beverage in the past month;
* be able to read English;
* reside in New Zealand;
* be a member of the online panel of "Research Now Survey Sampling International".

Exclusion Criteria:

* Participants not meeting the eligibility criteria will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 615 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2018-09-23 (Actual); Study Completion 2018-09-23 (Actual)

PRIMARY OUTCOMES:
Consumer online purchasing behaviour | Measured immediately after randomization
  Consumer online purchasing behaviour assessed on an 11-point Juster scale (where 1 = no chance/almost no chance and 11 = certain/practically certain

SECONDARY OUTCOMES:
Purchase behaviour | Measured immediately after randomization
  Number of alcoholic beverage(s) bought in the online shopping cart
Perceived and estimated energy content of displayed product | Measured at randomization
  Assessed using a seven-point scale ranging from "very low" to "very high" and the estimated energy content of the product
Perceived confidence in estimating energy content of displayed product | Measured immediately after randomization
  assessed using a seven-point scale ranging from "not confident at all" to "very confident"
Intention to consume displayed product | Measured immediately after randomization
  Assessed using a seven-point scale ranging from "would decrease consumption level" to "would increase consumption level"
Attitudes towards displayed product | Measured immediately after randomization
  On a seven-point rating scale participants will be asked whether they believe the displayed alcoholic product was expensive/cheap, unattractive/attractive, low quality/high quality, unhealthy/healthy, and taste bad/good.
Support for displayed label | Measured at randomization
  On a seven-point rating scale participants will be asked whether they would support the implementation of the displayed label
Attitudes towards alcohol | Measured immediately after randomization
  Assessed using the Scale for Measurement of Attitudes Towards Alcohol, a tool used to i) assess people's risk profile regarding the use of alcohol and ii) identify the factors that contribute to determining their attitudes

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Walker, PhD, Principal Investigator — University of Auckland, New Zealand
Locations (1):
- National Institute for Health Innovation, University of Auckland, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Walker N, McCormack J, Jiang, Y, Lang B, Ni Murchu C. (2018). Energy labelling for alcoholic beverages in New Zealand: Clinical trial. Phase 2 report: Wellington: Health Promotion Agency.
- [Result] Walker N, McCormack J, Jiang, Y, Lang B, Ni Murchu C. (2018). Energy labelling for alcoholic beverages in New Zealand: Consumer perceptions. Phase 1 report: Focus Groups. Wellington: Health Promotion Agency. ISBN:978-0-478-44956-3.